CLINICAL TRIAL: NCT04442100
Title: The Study of Biological Prosthetic Heart Valves With the "Easy Change" System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Konstantin A. Petlin, Ekaterina Alekseevna Kosovskikh, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Easy Change
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bioprosthesis (Experimental): prosthetics of heart valves with dentures "MedEng-Bio"
  Interventions: Procedure: valve prosthetics

INTERVENTIONS:
Procedure: valve prosthetics — prosthetics of heart valves with dentures "MedEng-Bio"

SUMMARY:
The study of new biological heart valves with the "easy change" system, including an assessment of the basic hemodynamic characteristics of the prosthesis, complications associated with valve implantation, and general mortality

DETAILED DESCRIPTION:
The study of new biological heart valves with the "easy change" system, including an assessment of the basic hemodynamic characteristics of the prosthesis, complications associated with valve implantation, and general mortality. Antithrombotic therapy after new biological valve prosthesis is studied. Transesophageal ultrasound is used for assessment of aortic strain, left ventricular strain, and 3D reconstruction of implanted bioprosthesis. The quality of life of patients is assessed using SF36 questionnaire. Heart failure after surgery is assessed by six-minute walking test and plasma BNP level.

ELIGIBILITY:
Inclusion Criteria:

1. aortic valve disease requiring surgical disease patients without symptoms with severe aortic stenosis - indexed area of the opening less than 0.5 cm2 / m2, average gradient more than 40 mm RT. Art;

   o patients who require coronary artery bypass grafting with moderate aortic stenosis - indexed area of the hole 0.5 - 1 cm2 / m2, the average gradient is more than 20 mm RT. Art., Regardless of symptoms;patients with symptoms of aortic stenosis, regardless of the severity of stenosis)
2. mitral valve disease requiring surgical disease

Exclusion Criteria:

1. the need for prosthetics of two or more valves
2. patients with a decrease in LVEF of less than 45%;
3. the presence of a competing disease or concomitant pathology that significantly affects the prognosis of quality of life or the likelihood of death
4. high pulmonary hypertension (SDJ above 60 mm Hg. Art.);
5. the diameter of the ascending aorta is more than 45 mm;
6. unwillingness of the patient to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
death | 10 years after surgery
  death from any cause
prosthetic complications | 10 years after surgery
  thromboembolism, infectious endocarditis, hemorrhage, structural valve degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Boris N. Kozlov, MD, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk, Tomsk Oblast, Russia